CLINICAL TRIAL: NCT03886337
Title: Evaluation of the Impact of Germicidal Light on Intraoperative S. Aureus Exposure
Brief Title: Impact of Germicidal Light
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started due to administrative reasons.
Sponsor: University of Iowa (Other)
Collaborators: Kenall Manufacturing (Other)
Responsible Party: Principal Investigator, Randy Loftus, Associate Professor of Anesthesia and Critical Care Medicine, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201901773
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Bacterial Transmission; S.Aureus Transmission; Operating Room Exposure to S. Aureus; 90-day Postoperative Surgical Site Infections, Superficial and Deep
Keywords: Germicidal lights; S. aureus; Transmission; Operating room S. aureus exposure
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): The control arm will be surgical care according to usual practice with usual ambient lighting
- Treatment Arm (Experimental): The treatment arm will include surgical care according to usual practice with germicidal ambient lighting
  Interventions: Device: Germicidal lighting

INTERVENTIONS:
Device: Germicidal lighting — Germicidal ambient lighting
  Arms: Treatment Arm

SUMMARY:
Visible light at 405nm has been shown to be germicidal. The hypothesis is that use of this light (Indigo-Clean Lights) in operating rooms will reduce S. aureus transmission occurring within and between patients and reduce surgical site infections (SSIs). Investigators will evaluate a case-control study where patients undergoing surgery with the lights are matched with patients undergoing surgery without germicidal lights.

DETAILED DESCRIPTION:
Operating room S. aureus exposure has been directly linked to postoperative infections and is therefore an important target for infection prevention. Visible light at 405nm has been shown to be germicidal. Investigators plan to install ambient, germicidal lighting (Indigo-Clean Lights) that uses this wavelength in 4 operating rooms. Patients will undergo surgery according to usual practice. Investigators will conduct a case-control study where patients undergoing surgery with the lights are matched with patients undergoing surgery without the germicidal lights. Patients will be matched by procedure then case duration then American Society of Anesthesiologists (ASA) physical status health classification. These patients will undergo infection surveillance. Infection surveillance will involve use of National Healthcare Safety Network (NHSN) checklists applied to patients who are positive for one or more of the initial screening criteria (elevated white blood cell count, fever (>38.4 degrees Celsius), office note documentation of infection, positive culture (sputum, blood, urine, wound, other body fluid), or anti-infective order within the 90 postoperative day period.

ELIGIBILITY:
Inclusion Criteria:

* Adult, at least 18 years old
* Adult patients undergoing orthopedic, cardiothoracic, gyn/onc, and neuro surgery and general anesthesia according to usual care with peripheral and/or central venous access.

Exclusion Criteria:

* Pediatric (<18 years old),
* Incarcerated, and/or
* Pregnant patients
* Undergoing surgery and/or without peripheral or central venous access.
* Undergoing surgery outside of the classifications above

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
S. aureus reservoir detection and/or epidemiologically-related transmission event in an OR observational unit. | Approximately 103 work days
  OR reservoirs will be surveyed for S. aureus isolation and epidemiologically-relatedness assessed

SECONDARY OUTCOMES:
90-day postoperative SSIs, superficial and/or deep. | 1.6 years
  surveillance of wound infections, superficial and deep
90-day HAIs (combined incidence of SSIs, respiratory, blood stream, catheter-associated urinary tract, and C. Difficile infections). | 1.6 years
  Surveillance of other healthcare-associated infections (HAIs)

CONTACTS AND LOCATIONS:
Overall Officials: Randy W. Loftus, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD related to the registered primary (S. aureus transmission dynamics) and secondary outcomes (healthcare-associated infections) will be shared freely with scientists who request them. The request process will require submission and review of a research proposal for data use by the PI (Loftus) and Indigo-Clean.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.

REFERENCES:
- [Background] Loftus RW, Dexter F, Robinson ADM. High-risk Staphylococcus aureus transmission in the operating room: A call for widespread improvements in perioperative hand hygiene and patient decolonization practices. Am J Infect Control. 2018 Oct;46(10):1134-1141. doi: 10.1016/j.ajic.2018.04.211. Epub 2018 Jun 12. PMID 29907449
- [Background] Loftus RW, Dexter F, Robinson ADM. Methicillin-resistant Staphylococcus aureus has greater risk of transmission in the operating room than methicillin-sensitive S aureus. Am J Infect Control. 2018 May;46(5):520-525. doi: 10.1016/j.ajic.2017.11.002. Epub 2018 Jan 4. PMID 29307750
- [Background] Loftus RW, Dexter F, Robinson ADM, Horswill AR. Desiccation tolerance is associated with Staphylococcus aureus hypertransmissibility, resistance and infection development in the operating room. J Hosp Infect. 2018 Nov;100(3):299-308. doi: 10.1016/j.jhin.2018.06.020. Epub 2018 Jun 30. PMID 29966756
- [Background] Magill SS, O'Leary E, Janelle SJ, Thompson DL, Dumyati G, Nadle J, Wilson LE, Kainer MA, Lynfield R, Greissman S, Ray SM, Beldavs Z, Gross C, Bamberg W, Sievers M, Concannon C, Buhr N, Warnke L, Maloney M, Ocampo V, Brooks J, Oyewumi T, Sharmin S, Richards K, Rainbow J, Samper M, Hancock EB, Leaptrot D, Scalise E, Badrun F, Phelps R, Edwards JR; Emerging Infections Program Hospital Prevalence Survey Team. Changes in Prevalence of Health Care-Associated Infections in U.S. Hospitals. N Engl J Med. 2018 Nov 1;379(18):1732-1744. doi: 10.1056/NEJMoa1801550. PMID 30380384
- [Background] Koff MD, Brown JR, Marshall EJ, O'Malley AJ, Jensen JT, Heard SO, Longtine K, O'Neill M, Longtine J, Houston D, Robison C, Moulton E, Patel HM, Loftus RW. Frequency of Hand Decontamination of Intraoperative Providers and Reduction of Postoperative Healthcare-Associated Infections: A Randomized Clinical Trial of a Novel Hand Hygiene System. Infect Control Hosp Epidemiol. 2016 Aug;37(8):888-895. doi: 10.1017/ice.2016.106. Epub 2016 Jun 7. PMID 27267310